CLINICAL TRIAL: NCT02221141
Title: Screening of Fabry Disease in Patients With Left Ventricular Hypertrophy Detected in Echocardiography
Status: Completed | Type: Observational
Sponsor: Laurence Gabriel (Other)
Responsible Party: Sponsor-Investigator, Laurence Gabriel, Dr Laurence GABRIEL, Centre Hospitalier Universitaire UCLouvain Namur
Organization: Centre Hospitalier Universitaire UCLouvain Namur (Other)
Other Study IDs: Fabry Disease Cardioscreening
Record Dates: First submitted 2014-08-18; First posted 2014-08-20 (Estimated); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Left Ventricular Hypertrophy
MeSH Terms: conditions — Hypertrophy, Left Ventricular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other

SUMMARY:
The purpose of this study is to determine the prevalence in Belgium of Fabry disease in patients with unexplained hypertrophic cardiomyopathy measured by echocardiography and to determine in Fabry patients which was the most frequently initial symptom.

Actually the early diagnosis is important because a treatment exists that can prevent future complications.

ELIGIBILITY:
Inclusion Criteria:

* unexplained left ventricular hypertrophy

Exclusion Criteria:

* isolated septal hypertrophy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with left ventricular hypertrophy
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2013-12; Primary Completion 2021-04 (Actual); Study Completion 2021-04 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with left ventricular hypertrophy who have Fabry Disease mutation | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dinant-Godinne, Yvoir, Belgium